CLINICAL TRIAL: NCT05258188
Title: Study Comparing the Effectiveness of Ergon Instruments-Assisted Soft Tissue Mobilization Techniques With Compressive Myofascial Release for Plantar Fasciitis: A Randomised Clinical Trial
Brief Title: Comparison of Ergon Instruments-Assisted Soft Tissue Mobilization With Compressive Myofascial Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-FSD-00266
Record Dates: First submitted 2022-02-20; First posted 2022-02-28 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Plantar Fasciitis
Keywords: Plantar Fascitis; Randomized Control Trial; Myofascial Release; Soft Tissue Mobilization; Ergon Instruments; Comparison
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Our study will be single-blinded, outcome assessor-blinded. The assessor will be blinded to avoid being biased during the outcome assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instrument-assisted Soft Tissue Mobilization (Experimental): 1. Warm-up will be performed for 10 to 15 minutes by light jogging, elliptical machine, stationary cycle or an upper body ergometer
  2. Instrument-assisted Soft Tissue Mobilization , will be applied at 30 to 60 degrees angle for 40 to 120 seconds
  3. Stretching, for 30 seconds (3 rep)
  4. Strengthening exercises, high repetitions with low intensity exercise
  5. Cryotherapy for 10 to 20 min
  Interventions: Other: Instrument-assisted Soft Tissue Mobilization
- Compressive Myofascial Release Technique (Experimental): Compressive myofascial release technique will be applied 5 minutes, after a warmup of 10 to 15 minutes.
  Interventions: Other: Compressive Myofascial Release Technique

INTERVENTIONS:
Other: Instrument-assisted Soft Tissue Mobilization — Instrument-assisted soft tissue mobilization is used for a mechanical benefit for the therapist providing deeper approach and braces remodeling of connective tissues through dissolution of extravagant fibrosis, while provoking repair and reconstructing forwarded by the recruitment of fibroblast.
  Arms: Instrument-assisted Soft Tissue Mobilization
Other: Compressive Myofascial Release Technique — Compressive Myofascial Release Technique is a technique of soft tissue stretching that uses compression and sustained myofascial stretches to create a releasing force in the targeted area
  Arms: Compressive Myofascial Release Technique

SUMMARY:
The objective of this study is to investigate the effects of Virtual Reality and Motor Imagery along with Routine Physical Therapy in motor function and balance in patients with Parkinson disease.

DETAILED DESCRIPTION:
This randomized control trial is the single blinded, single centered study. Standard Protocol Items: Recommendations for Interventional Trials guidelines are used as study protocol. Sixty three patients of Parkinson Disease (Modified Hoehn and Yahr stages I-III) will randomly allocate into three groups.

Group A will be given a 60 min session of Virtual Reality along with Routine Physical Therapy.

Group B will be given a 60 min session of Motor Imagery along with Routine Physical Therapy.

Group C will be given a 40 min session of Routine Physical Therapy and after a short period of rest,20 min for walking and cycling.

These treatment sessions will be given to each group at every alternative day (3 days per week) for 12 weeks.

Outcome measures are

1. Berg Balance Scale
2. Activities Specific Balance Confidence Scale
3. The Unified Parkinson Disease Rating Scale (part III) The Assessments will be recorded at baseline, at 6th and 12th weeks of therapy, and after one month of discontinuation of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Inability to achieve 20 degrees of active dorsiflexion,
* Heel pain,
* Mid foot pain,
* Heal swelling,
* Mid foot swelling,
* Achilles' tendon tightness diagnosed on the base of Windlass test

Exclusion Criteria:

* Recent foot injury,
* Fracture,
* Infections,
* Surgical procedures,
* Tendon injury,
* Hypermobility,
* Neuromuscular disorders,
* Impaired sensation,
* Open sores,
* Skin disease,
* Active deep vein thrombosis or thrombophlebitis,
* Bruises,
* Varicose veins,
* Burn scars

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Range of Motion | 12th Week
  Goniometer has been the most widely used tool for measuring joint range of motion. To ensure reliable measurement, standardized, specific positions and landmarks are used to measure each joint movement.
Visual Analogue Scale | 12th Week
  The Visual Analog Scale is a 10 cm line with anchor statements on the left, no pain and on the right, extreme pain.
Foot and Ankle Disability Index | 12th Week
  The Foot and Ankle Disability Index has 26 items. Each item is scored from 0; unable to do, to 4; no difficulty at all. The Foot and Ankle Disability Index has a total point value of 104 points.
Foot and Ankle Ability Measure | 12th Week
  The Foot and Ankle Ability Measure (FAAM) is a self-report outcome instrument/questionaire developed to assess physical function for individuals with foot and ankle related impairments. 8-item Sports Subscale.
  Each item is scored on a 5-point Likert scale (4 to 0) from 'no difficulty at all' to 'unable to do'. Item score totals, which range from 0 to 84 for the ADL subscale and 0 to 32 for the Sports subscale, were transformed to percentage scores. Higher scores represent higher levels of function for each subscale, with 100% representing no dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No